CLINICAL TRIAL: NCT00093002
Title: A Randomized, Open-Label, Multicenter, Phase II Study Comparing the Effects on Proliferation and the Efficacy and Tolerability of Fulvestrant (FASLODEX®) 500 mg With Fulvestrant (FASLODEX®) 250 mg When Given as Neoadjuvant Treatment in Postmenopausal Women With Estrogen Receptor Positive Breast Cancer (T2, 3, 4b, N0-3, M0).
Brief Title: Fulvestrant (FASLODEX™) as a Treatment in Postmenopausal Women With Estrogen Receptor Positive Breast Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 9238IL/0065; D6997C00003
Record Dates: First submitted 2004-09-28; First posted 2004-09-29 (Estimated); Last update posted 2008-06-12 (Estimated); Status verified 2008-06

CONDITIONS: Breast Cancer
Keywords: Early Breast Cancer; neoadjuvant therapy; hormonal treatment; newly diagnosed breast cancer; Estrogen Receptor Positive Breast Cancer; treatment naïve; neoadjuvant treatment; neoadjuvant setting; invasive breast cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Fulvestrant

ARMS (2):
- 1 (Experimental): 250 mg fulvestrant
  Interventions: Drug: Fulvestrant
- 2 (Experimental): 500 mg fulvestrant
  Interventions: Drug: Fulvestrant

INTERVENTIONS:
Drug: Fulvestrant — 250 mg & 500 mg intramuscular injection
  Other Names: FASLODEX™; ZD9238

SUMMARY:
The purpose of this study is to evaluate fulvestrant in the preliminary stage of breast cancer treatment and assess the relationship between dose, exposure, degree of reduction in tumor markers, and efficacy in postmenopausal women with estrogen receptor positive disease.

ELIGIBILITY:
Inclusion Criteria:

* Postmenopausal women defined as women who have stopped having menstrual periods
* Written informed consent to participate in the trial
* Biopsy confirmation of invasive breast cancer
* Evidence of hormone sensitivity
* Willingness to undergo biopsies

Exclusion Criteria:

* Any previous treatment for breast cancer
* Unwillingness to stop taking any drug known to affect sex hormonal status or a patient in which it would be inappropriate to stop.
* Any severe concurrent condition that would preclude surgery or that would jeopardize compliance with the study, e.g., uncontrolled cardiac disease or uncontrolled diabetes mellitus
* The presence of more than one primary tumor
* History of hypersensitivity to castor oil
* History of known bleeding disorders

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 179 (Actual)
Dates: Start 2004-06; Study Completion 2007-07 (Actual)

PRIMARY OUTCOMES:
Anti-proliferative effect after 4 weeks of treatment.

SECONDARY OUTCOMES:
Safety, tolerability, tumor response and pharmacokinetics after 4 weeks of treatment.

CONTACTS AND LOCATIONS:
Overall Officials: AstraZeneca Faslodex Medical Science Director, MD, Study Director — AstraZeneca
Locations (31):
- United States (7):
  - Research Site, Little Rock, Arkansas
  - Research Site, Boston, Massachusetts
  - Research Site, Winchester, Massachusetts
  - Research Site, Albuquerque, New Mexico
  - Research Site, Hershey, Pennsylvania
  - Research Site, Nashville, Tennessee
  - Research Site, Laredo, Texas
- Austria (3):
  - Research Site, Innsbruck
  - Research Site, Salzburg
  - Research Site, Vienna
- Brazil (7):
  - Research Site, Barretos
  - Research Site, Florianópolis
  - Research Site, Goiamia
  - Research Site, Porto Alegre
  - Research Site, Rio de Janeiro
  - Research Site, Santo André
  - Research Site, São Paulo
- Germany (5):
  - Research Site, Berlin
  - Research Site, Hanover
  - Research Site, Magdeburg
  - Research Site, München
  - Research Site, Rostock
- India (5):
  - Research Site, Bangalore
  - Research Site, Hyderabaad
  - Research Site, New Delhi
  - Research Site, Pune
  - Research Site, Trivandrum
- United Kingdom (4):
  - Research Site, Birmingham
  - Research Site, Bournemouth
  - Research Site, Dundee
  - Research Site, Edinburgh

REFERENCES:
- See also: Medline Plus - Information on Breast Cancer — http://www.nlm.nih.gov/medlineplus/breastcancer.html
- See also: Breastcancer.org — http://www.breastcancer.org/